CLINICAL TRIAL: NCT06985550
Title: Effect of Adding Additional Elastic Band Resistance Training to Waltz Dance on Dyslipidemia in Middle-aged and Elderly Women: a Randomized Controlled Trial
Acronym: MEP&DL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Principal Investigator, Jiedan Luo, PHD, Gdansk University of Physical Education and Sport
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWFiS/2025_4_JL
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Dyslipaemia
Keywords: Dyslipaemia; Multicomponent Exercise; Waltz
MeSH Terms: interventions — Activities of Daily Living

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants in this group will participate in a 12-week multi-component exercise program, three times a week for 90 minutes each time. Each session includes a 5-minute warm-up, 50 minutes of waltz dancing (learning and practicing steps), 30 minutes of resistance band exercises (1-3 sets of 8-16 repetitions at 10-20 grams of maximum resting resistance), and 5 minutes of cool-down stretching. Exercise intensity will gradually increase from 50% to 75% of maximum heart rate (HRmax) (RPE 10-13, METs 2.0-6.0). The program aims to improve lipid profile, body composition, cardiovascular health, balance, mental health, and cognitive function in women aged 65 and under with dyslipidemia.
  Interventions: Behavioral: Multicomponent Exercise
- Control group (Other): Only daily activities are included.
  Interventions: Other: daily activity

INTERVENTIONS:
Behavioral: Multicomponent Exercise — Participants in this group will participate in a 12-week multi-component exercise program, three times a week for 90 minutes each time. Each session includes a 5-minute warm-up, 50 minutes of waltz dancing (learning and practicing steps), 30 minutes of resistance band exercises (1-3 sets of 8-16 repetitions at 10-20 grams of maximum resting resistance), and 5 minutes of cool-down stretching. Exercise intensity will gradually increase from 50% to 75% of maximum heart rate (HRmax) (RPE 10-13, METs 2.0-6.0). The program aims to improve lipid profile, body composition, cardiovascular health, balance, mental health, and cognitive function in women aged 65 and under with dyslipidemia.
  Arms: Exercise group
Other: daily activity — Only daily activities are included.
  Arms: Control group

SUMMARY:
Brief Summary:

This clinical trial aims to evaluate whether a 12-week multi-component exercise program (combining waltz, resistance training, and agility training) can improve the physical, psychological, and cognitive function of women aged 65 and under with dyslipidemia. Key research questions include: Does this intervention lower lipid levels (e.g., total cholesterol, triglycerides) and improve body composition (e.g., body fat percentage, lean muscle mass)? Compared to a non-exercise control group, does this intervention enhance cardiovascular health, balance, mental health, and cognitive function? Researchers will compare outcomes in the exercise intervention group and the non-exercise control group to assess the effectiveness of the program. Study Procedure: Participants will: attend supervised exercise classes three times a week for 12 weeks (approximately 90 minutes per class). The program includes: - Waltz training (basic steps and choreographed dance movements), - Resistance band exercises (targeting major muscle groups), - Agility and balance training modules. Pre- and post-intervention assessments will include: - Lipid analysis, - Body composition analysis, - Cardiovascular health and balance tests, - Standardized mental health and cognitive assessments.

ELIGIBILITY:
Inclusion Criteria

1. Female, aged 45 to 65 years
2. Diagnosis of dyslipidemia defined according to the National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) criteria, meeting at least one of the following:

   Total cholesterol ≥ 200 mg/dL Low-density lipoprotein cholesterol ≥ 130 mg/dL Triglycerides ≥ 150 mg/dL High-density lipoprotein cholesterol < 50 mg/dL
3. Not taking lipid-lowering medications, or on a stable lipid-lowering regimen for at least 3 months prior to enrollment with no anticipated changes during the study period
4. Medically cleared to participate in moderate-intensity aerobic and resistance exercise according to American College of Sports Medicine (ACSM) guidelines
5. Able and willing to participate in a 12-week supervised exercise intervention
6. Provided written informed consent

Exclusion Criteria

1. History of major cardiovascular events, including myocardial infarction, stroke, or unstable angina
2. Diagnosed diabetes with poor glycemic control
3. Serious metabolic or endocrine diseases known to affect lipid metabolism (e.g., uncontrolled thyroid disease)
4. Serious musculoskeletal, neurological, or orthopedic conditions that may limit safe participation in sports
5. Participated in a structured exercise program more than 2 times per week in the past 6 months
6. Current hormone replacement therapy or other medications known to significantly affect lipid metabolism
7. Cognitive impairment or psychiatric illness that may interfere with study participation or adherence
8. Any other medical condition that was deemed by the investigators to compromise the safety of the participants or the integrity of the data

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 60 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol (TC) Level | From baseline through the end of the 12-week intervention period
  Total cholesterol will be measured in fasting venous blood samples (12-hour fast) using an enzymatic colorimetric method with a clinical chemistry analyzer. The result will be reported in mg/dL. Total cholesterol refers to the overall amount of cholesterol in the blood, which includes LDL-C and HDL-C. High levels are associated with increased cardiovascular risk. Blood samples will be collected at baseline and at the end of the 12-week intervention.
Triglycerides (TG) Level | From baseline through the end of the 12-week intervention period
  Triglyceride levels will be measured from fasting venous blood samples (12-hour fast) using enzymatic assays with a clinical chemistry analyzer. The result will be reported in mg/dL. Triglycerides are a type of fat found in the blood. Elevated levels are associated with metabolic syndrome and increased risk of heart disease. Blood samples will be collected at baseline and at 12 weeks post-intervention.
High-Density Lipoprotein Cholesterol (HDL-C) Level | From baseline through the end of the 12-week intervention period
  HDL-C will be measured from fasting venous blood samples using direct enzymatic assays. HDL-C is often referred to as "good" cholesterol because it helps remove other forms of cholesterol from the bloodstream. Low levels are a risk factor for cardiovascular disease. The result will be reported in mg/dL and assessed at baseline and after the 12-week program.
Low-Density Lipoprotein Cholesterol (LDL-C) Level | From baseline through the end of the 12-week intervention period
  LDL-C will be measured using the Friedewald equation or direct measurement (depending on TG level) from fasting venous blood samples. LDL-C is known as "bad" cholesterol because it contributes to plaque buildup in arteries. The result will be reported in mg/dL. Blood samples will be taken at baseline and after the 12-week exercise intervention.

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure (SBP, DBP) | From baseline through the end of the 12-week intervention period
  Resting systolic and diastolic blood pressure will be measured using a validated automatic digital blood pressure monitor (e.g., Omron HEM-907). Participants will be seated quietly for at least 5 minutes prior to measurement. Three readings will be taken at 1-minute intervals on the non-dominant arm, and the average of the last two will be recorded. Blood pressure is expressed in mmHg and interpreted according to international hypertension guidelines.
Cardiorespiratory Fitness (Estimated VO₂max via 6-Minute Walk Test) | From baseline through the end of the 12-week intervention period
  Cardiorespiratory fitness will be estimated using the 6-Minute Walk Test (6MWT), a validated submaximal field test. Participants will be instructed to walk at their fastest safe pace along a 30-meter corridor for 6 minutes. Total distance covered will be used to estimate VO₂max using validated predictive equations adjusted for age and sex. This measure reflects aerobic capacity and endurance.
Vascular Function (Pulse Wave Velocity [PWV], Ankle-Brachial Index [ABI]) | From baseline through the end of the 12-week intervention period
  Arterial stiffness and peripheral vascular health will be assessed using a validated vascular testing device (e.g., VaSera VS-1500 or equivalent). Pulse Wave Velocity (PWV) measures the speed of arterial pulse propagation and is a marker of arterial stiffness. Ankle-Brachial Index (ABI) is calculated by dividing the systolic blood pressure at the ankle by that at the brachial artery. Both are non-invasive and widely used indicators of cardiovascular health.
Body Composition | From baseline through the end of the 12-week intervention period
  Body composition will be assessed using a validated bioelectrical impedance analysis device (e.g., InBody 720), including body fat percentage, body fat mass, lean body mass, skeletal muscle mass, and body mass index (BMI). Participants will be measured barefoot and in light clothing after an overnight fast, following standard procedures recommended by the manufacturer.
Bone Mineral Density (BMD) | From baseline through the end of the 12-week intervention period
  Bone mineral density will be evaluated using an ultrasound bone densitometer (e.g., Sahara Clinical Bone Sonometer), measuring the calcaneal bone (heel). The test is non-invasive, and results will be recorded as T-scores according to WHO criteria.
Static Balance | From baseline through the end of the 12-week intervention period
  Static balance will be assessed using the single-leg stance test with eyes closed. The maximum duration (in seconds) the participant can stand unassisted on one leg without touching the ground with the lifted foot will be recorded, up to 60 seconds. Three trials will be conducted and the best result recorded.
Dynamic Balance | From baseline through the end of the 12-week intervention period
  Dynamic balance will be measured using the Biodex Balance System SD, performing the Limits of Stability (LOS) test protocol. Participants will stand on a movable platform and shift their center of gravity to targets displayed on a screen. Scores will reflect directional control and stability performance.

OTHER OUTCOMES:
Anxiety - Generalized Anxiety Disorder 7-item scale (GAD-7) | From baseline through the end of the 12-week intervention period
  Anxiety symptoms will be evaluated using the GAD-7, a validated self-report scale assessing the frequency of anxiety-related symptoms over the past two weeks. Each item is scored from 0 ("not at all") to 3 ("nearly every day"), with a total score range of 0-21. Higher scores indicate greater anxiety severity.
Depression - Patient Health Questionnaire-9 (PHQ-9) | From baseline through the end of the 12-week intervention period
  Depressive symptoms will be assessed using the PHQ-9, a widely used 9-item self-report measure based on DSM-IV criteria. Participants rate the frequency of symptoms over the past two weeks. Scores range from 0 to 27, with higher scores indicating more severe depression.
Mood State - Profile of Mood States (POMS) | From baseline through the end of the 12-week intervention period
  Mood state will be measured using the Profile of Mood States (POMS), a 65-item self-report questionnaire that evaluates six mood dimensions: tension, depression, anger, vigor, fatigue, and confusion. Scores are combined to generate a total mood disturbance score.
Exercise Motivation - Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3) | From baseline through the end of the 12-week intervention period
  Exercise motivation will be measured using the BREQ-3, which evaluates different types of motivational regulation along the self-determination continuum, including intrinsic motivation, identified regulation, introjected regulation, external regulation, and amotivation. The scale uses a 5-point Likert response format.
Cognitive Function - Montreal Cognitive Assessment (MoCA) | From baseline through the end of the 12-week intervention period
  Global cognitive function will be assessed using the MoCA, a validated screening tool for mild cognitive impairment. The MoCA evaluates attention, memory, language, executive function, visuospatial skills, and orientation. The maximum score is 30, with scores below 26 indicating possible cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education, Sichuan Normal University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The dataset will remain confidential in accordance with ethical and regulatory requirements to protect participant privacy.